CLINICAL TRIAL: NCT02470234
Title: A Pharmacokinetic Study of Aptensio XR® (Methylphenidate Hydrochloride (HCl) Extended-release) Capsules in Male or Female Pre-School Children 4 to Under 6 Years of Age With Attention Deficit Hyperactivity Disorder (ADHD) in Fed Condition
Brief Title: Pharmacokinetic Study of Methylphenidate HCl Extended-Release Capsules in Children 4 to Under 6 Years of Age With ADHD
Acronym: PK003
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RP-BP-PK003
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; Children; Pharmacokinetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methylphenidate HCl ER Capsules, 10 mg (Experimental): Methylphenidate Hydrochloride Extended Release Capsules, 10 mg. Active drug, administered once
  Interventions: Drug: Methylphenidate HCl ER Capsules, 10 mg
- Methylphenidate HCl ER Capsules, 15 mg (Experimental): Methylphenidate Hydrochloride Extended Release Capsules, 15 mg. Active drug, administered once
  Interventions: Drug: Methylphenidate HCl ER Capsules, 15 mg
- Methylphenidate HCl ER Capsules, 20 mg (Experimental): Methylphenidate Hydrochloride Extended Release Capsules, 20 mg. Active drug, administered once
  Interventions: Drug: Methylphenidate HCl ER Capsules, 20 mg

INTERVENTIONS:
Drug: Methylphenidate HCl ER Capsules, 10 mg — Methylphenidate Hydrochloride Extended-Release Capsules, 10 mg administered once daily in the morning
  Other Names: Aptensio XR®, 10 mg
  Arms: Methylphenidate HCl ER Capsules, 10 mg
Drug: Methylphenidate HCl ER Capsules, 15 mg — Methylphenidate Hydrochloride Extended-Release Capsules, 15 mg administered once daily in the morning
  Other Names: Aptensio XR®, 15 mg
  Arms: Methylphenidate HCl ER Capsules, 15 mg
Drug: Methylphenidate HCl ER Capsules, 20 mg — Methylphenidate Hydrochloride Extended-Release Capsules, 20 mg administered once daily in the morning
  Other Names: Aptensio XR®, 20 mg
  Arms: Methylphenidate HCl ER Capsules, 20 mg

SUMMARY:
To assess the pharmacokinetics of a single dose of Aptensio XR® (methylphenidate hydrochloride extended-release) capsules under fed conditions in male or female children 4 to under 6 years of age with ADHD.

DETAILED DESCRIPTION:
This will be a multi-center, open-label, single-dose, study to assess the pharmacokinetics of Aptensio XR® (methylphenidate hydrochloride extended-release) capsules in male and female children 4 to under 6 years of age with ADHD in fed condition.

Screening Procedures: After obtaining written informed consent from parents, subjects will undergo a complete medical and medication history, demographic data (including sex, age, race, ethnicity, body weight (kg), height (cm), Body Mass Index (BMI) (kg/m2), physical examination, vital signs evaluation (sitting blood pressure, pulse rate, respiration rate, temperature and pulse oximetry), resting 12-lead electrocardiogram (ECG), clinical laboratory tests and concomitant medication within 28 days prior to receiving study drug. On Day 1: subjects will receive a single oral dose of Aptensio XR®.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or female between the ages of 4 and under 6 years old.
2. Patient has a history consistent with ADHD, meets the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for ADHD, inattentive, hyperactivity or combined.
3. Patient must meet criteria for ADHD diagnosis on Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime (KSADS-PL) and clinical interview by experienced clinician; symptoms must have been present for at least 6 months.
4. Subject has had prior behavioral treatment or subject's symptoms are severe enough to warrant treatment without prior behavioral treatment, and patient is on a stable dose of either immediate-release or extended-release methylphenidate.
5. Subject must have age- and sex-adjusted ratings of ≥ 90th percentile Total Score on the Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Preschool Version, a Clinical Global Impressions -Severity Score of ≥4 and a Child Global Assessment Scale rating of <65 after methylphenidate washout and prior to obtaining pharmacokinetic samples. Ratings may be completed via telephone on day-1.
6. Parents or guardians of patients must have the ability to read and understand the language in which the Informed Consent is written and are mentally and physically competent to provide written informed consents for their child.
7. Patient and/or parent are/is able to understand English in order to provide assent and is otherwise able to comply with the study protocol.

Exclusion Criteria:

1. Patient has allergy to methylphenidate or amphetamines, or history of serious adverse reaction to methylphenidate.
2. Patient has a history of tension, agitation, glaucoma, thyrotoxicosis, tachyarrhythmias or severe angina pectoris or patient with serious or unstable medical illness such as asthma, diabetes or seizures.
3. A history of motor or vocal tics or Tourette's syndrome
4. Patient is receiving monoamine oxidase inhibitors, anticonvulsants (phenobarbital, phenytoin, primidone), coumarin anticoagulants, presser agents, guanethidine, tricyclic antidepressants (imipramine, desipramine, selective serotonin inhibitors (SSRIs), or herbal remedies (e.g., melatonin).
5. Patient has serious hypertension.
6. Patient has a history of disorders of the sensory organs, particularly deafness, severe or profound retardation.
7. Patient has any other unstable psychiatric condition requiring treatment.
8. Patient is at risk for substance abuse.
9. Evidence of current physical, sexual, or emotional abuse
10. Living with anyone who currently abuses stimulants or cocaine
11. History of bipolar disorder in both biological parents

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-07-30 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akwete Adjei, Ph.D., Study Director — Rhodes Pharmaceuticals, L.P.
Locations (2):
- United States (2):
  - Qps-Mra, Llc, South Miami, Florida
  - Duke Psychiatry and Behavioral Sciences, Duke University School of Medicine, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adjei AL, Chaudhary I, Kollins SH, Padilla A. A Pharmacokinetic Study of Methylphenidate Hydrochloride Multilayer Extended-Release Capsules (Aptensio XR(R)) in Preschool-Aged Children with Attention-Deficit/Hyperactivity Disorder. Paediatr Drugs. 2020 Oct;22(5):561-570. doi: 10.1007/s40272-020-00409-z. PMID 32776159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was a parallel design study, where subjects were recruited from July 02, 2016 - July 19, 2017. Eligible subjects received one capsule of Methylphenidate HCl ER (10, 15, 20, 30, or 40 mg) on only one of the 3 dosing days depending on number of subjects recruited up each particular dosing day. Only 1 site was able to recruit subjects.
Groups:
- Methylphenidate HCl ER 10 mg: Subjects received a single dose of Methylphenidate HCl ER 10 mg . This dose was equivalent to their current total daily methylphenidate dose.
- Methylphenidate HCl ER 15 mg: Subjects received a single dose of Methylphenidate HCl ER 15 mg . This dose was equivalent to their current total daily methylphenidate dose.
- Methylphenidate HCl ER 20 mg: Subjects received a single dose of Methylphenidate HCl ER 20 mg . This dose was equivalent to their current total daily methylphenidate dose.
Period: Overall Study
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Started | 5 | 3 | 2
Completed | 5 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Methylphenidate HCl ER 10 mg: Subjects received a single dose of Methylphenidate HCl ER 10 mg
- Methylphenidate HCl ER 15 mg: Subjects received a single dose of Methylphenidate HCl ER 15 mg
- Methylphenidate HCl ER 20 mg: Subjects received a single dose of Methylphenidate HCl ER 20 mg
- Total: Total of all reporting groups
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg | Total
Number analyzed (Participants) | 5 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: Months] | 61.0 (8.03) | 63.3 (5.51) | 70.5 (0.71) | 63.6 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 4 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 4 | 2 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 6
  White | 0 | 1 | 1 | 2
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 15.3 (0.55) | 15.3 (0.98) | 15.3 (2.26) | 15.3 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Methylphenidate HCl ER 10 mg: Active drug, administered once
  Methylphenidate HCl ER 10 mg Capsule: Methylphenidate Hydrochloride Extended-Release Capsules single dose administered in the morning under fed conditions
- Methylphenidate HCl ER 15 mg; Methylphenidate HCl ER 20 mg: Active drug, administered once
  Methylphenidate HCl ER 15 mg Capsule: Methylphenidate Hydrochloride Extended-Release Capsules single dose administered in the morning under fed conditions
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 5 | 3 | 2
ng/mL | 8.07 (1.702) | 10.09 (0.620) | 15.45 (1.061)

2. Primary Outcome: AUC(0-t)
Description: Area under the plasma concentration versus time curve (calculated to the last measurable observation).
  AUC: Area Under the Curve
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Methylphenidate HCl ER 20 mg: Active drug, administered once
  Methylphenidate HCl ER 20 mg Capsule: Methylphenidate Hydrochloride Extended-Release Capsules single dose administered in the morning under fed conditions.
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 5 | 3 | 2
ng*hr/mL | 89.18 (25.047) | 118.49 (18.211) | 155.95 (35.209)

3. Primary Outcome: AUC(0-inf)
Description: Area under the plasma concentration versus time curve, extrapolated to infinity.
  AUC: Area Under the Curve
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per protocol. (n=1) Standard Deviation was not estimable.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 3 | 1 | 1
ng*hr/mL | 105.26 (21.831) | 140.68 (0) | 144.26 (0)

4. Primary Outcome: AUC/D
Description: Dose-normalized AUC0-t. AUC: Area Under the Curve
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol.
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 5 | 3 | 2
ng*hr/mL/mg | 8.92 (2.505) | 7.90 (1.214) | 7.80 (1.760)

5. Primary Outcome: CL/F
Description: Apparent clearance. CL: Clearance
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per protocol. (n=1) Standard Deviation was not estimable.
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- Methylphenidate HCl ER 20 mg Capsule: Active drug, administered once
  Methylphenidate HCl ER 20 mg Capsule: Methylphenidate Hydrochloride Extended-Release Capsules single dose administered in the morning under fed conditions.
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg Capsule
Number analyzed (Participants) | 3 | 1 | 1
L/h | 97.51 (18.095) | 106.63 (0) | 138.64 (0)

6. Primary Outcome: V(Dss)/F
Description: Volume of distribution
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per protocol. (n=1) Standard Deviation was not estimable.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 3 | 1 | 1
L | 682.49 (182.605) | 1952.17 (0) | 1396.96 (0)

7. Primary Outcome: Cmax/Dose
Description: Dose-normalized Cmax
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 5 | 3 | 2
ng/mL/mg | 0.81 (0.170) | 0.67 (0.041) | 0.77 (0.053)

8. Secondary Outcome: Tmax
Description: Time to peak plasma concentration
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol
Measure: Median (Full Range); unit: h
Groups:
- Methylphenidate HCl ER 10 mg: Active drug, administered once
  Methylphenidate HCl ER 10 mg Capsule: Methylphenidate Hydrochloride Extended-Release Capsules single dose administered in the morning under fed conditions.
  .
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 5 | 3 | 2
h | 2.0 [1.0 to 3.0] | 3.0 [3.0 to 12.0] | 2.0 [2.0 to 2.0]

9. Secondary Outcome: T1/2
Description: Elimination half-life
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol. (n=1) Standard Deviation was not estimable.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 3 | 1 | 1
h | 4.80 (0.466) | 12.69 (0) | 6.98 (0)

10. Secondary Outcome: Kel
Description: Terminal elimination constant
Time Frame: Day 1 at time 0 (within 30-60 minutes pre-dose) and 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: Per Protocol. (n=1) Standard Deviation was not estimable
Measure: Mean (Standard Deviation); unit: h-1
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
Number analyzed (Participants) | 3 | 1 | 1
h-1 | 0.15 (0.015) | 0.05 (0) | 0.10 (0)

ADVERSE EVENTS:
Time Frame: From check in until 24 hours post dose
Description: Definitions for SAEs and AEs do not differ from ClinicalTrials.gov definitions
Arm/Group | Methylphenidate HCl ER 10 mg | Methylphenidate HCl ER 15 mg | Methylphenidate HCl ER 20 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/5 | 0/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate HCl ER 10 mg (N=5) | Methylphenidate HCl ER 15 mg (N=3) | Methylphenidate HCl ER 20 mg (N=2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Not Related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT02470234/Prot_SAP_000.pdf